CLINICAL TRIAL: NCT02705677
Title: Biobanking of Rett Syndrome and Related Disorders Protocol
Brief Title: Biobanking of Rett Syndrome and Related Disorders
Status: Completed | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Center for Advancing Translational Sciences (NCATS) (NIH); Office of Rare Diseases (ORD) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Alan Percy, Principal Investigator, University of Alabama at Birmingham
Other Study IDs: RDCRN # 5213; U54HD061222 (NIH)
Record Dates: First submitted 2015-11-22; First posted 2016-03-10 (Estimated); Last update posted 2021-08-05 (Actual); Status verified 2021-08

CONDITIONS: Rett Syndrome; MECP2 Duplication; CDKL5; FOXG1 Disorders
MeSH Terms: conditions — Rett Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA and RNA from blood, plasma, hair follicles, skin biopsies
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Rett syndrome: This is a biobanking project for individuals with mutations in MECP2 or meeting diagnostic criteria for classic (typical) or variant (atypical) Rett syndrome in order to identify other genetic factors such as X-chromosome inactivation or genetic background that may explain the variations noted in these individuals, including those with the same MECP2 mutation. No interventions are anticipated.
- MECP2 Duplication disorder: This is a biobanking project for individuals with MECP2 duplications to understand the difference in the size of the duplication and the potential impact of other genes in the duplicated segment. No interventions are anticipated.
- Rett-related disorders: CDKL5, FOXG1: This is a biobanking project for individuals with mutations in MECP2, CDKL5, and FOXG1 to understand the interplay of mutations in these individuals and the resultant phenotypic expression; for example, individuals with mutations in MECP2 but not meeting diagnostic criteria for Rett syndrome or individuals with mutations in CDKL5 or FOXG1 who may or may not meet diagnostic criteria for atypical Rett syndrome. No interventions are anticipated.

SUMMARY:
The overarching purpose of this study is to advance understanding of the natural history of Rett syndrome (RTT), MECP2-duplication disorder (MECP2 Dup), RTT-related disorders including CDKL5, FOXG1, and individuals with MECP2 mutations who do not have RTT. Although all these disorders are the result of specific genetic changes, there remains broad clinical variation that is not entirely accounted for by known biological factors. Additionally, clinical investigators currently do not have any biomarkers of disease status, clinical severity, or responsiveness to therapeutic intervention. To address these issues, biological materials (DNA, RNA, plasma, cell lines) will be collected from affected individuals and in some cases from unaffected family members, initial evaluation performed to identify additional biological factors contributing to disease severity, and these materials will be stored for future characterization.

DETAILED DESCRIPTION:
At the present time, effective treatments for RTT, MECP2 Dup, or Rett-related disorders are lacking. Investigators have made substantial progress in RTT over the past eleven years such that this study represents a narrowing of focus to mutations or duplications of the MECP2 gene and related disorders, including those with phenotypic overlap. Understanding of RTT has advanced remarkably well through the Rett Syndrome Natural History Clinical Protocol (NHS) and correspondingly advancement in the basic science realm has moved forward with equivalent success. Thus, progress in clinical and basic science has led to the establishment of clinical trials and other translational studies that hold promise for additional clinical trials in future. In the process, however, investigators became aware of additional MECP2- and RTT-related disorders that were unknown at the time the original proposal was conceived and further were impressed by the substantial clinical variability in individuals with RTT that cannot be explained by differences in mutations alone. In fact, variability among individuals with identical mutations has led investigators to search for additional explanations. At the time of the initial application (2002), just three years after the identification of the gene, MECP2, as the molecular link to RTT, investigators were not aware of the variation in clinical disorders related to MECP2 mutations or to the related but quite different MECP2 Dup. Each disorder is characterized by significant neurodevelopmental features related either to alterations in the MECP2 gene or related to phenotypes closely resembling those seen in individuals with RTT. Further, the phenotypic overlap with RTT due to mutations in CDKL5 and FOXG1 was also unexplored. The investigators propose in this new study to build on the substantial progress made in understanding both classic and variant RTT and to add these related disorders, MECP2 Dup and the Rett-related disorders including CDKL5, FOXG1, and individuals with MECP2 mutations who do not have RTT. In conjunction with the longitudinal clinical assessment performed via the natural history component, investigators will systematically collect from all willing participant's blood and isolate plasma, DNA, and RNA. All participants in the Natural History Study will be asked to contribute samples at the initial visit, whereas samples will be collected repeatedly on a subset of participants in order to look for changes over time. In order to identify factors that distinguish between affected and unaffected individuals, as well as to have the potential to characterize the heritability and potential consequences of genetic changes in families, samples will be collected from unaffected family members. Additionally, on a subset of individuals chosen because of unique clinical features skin biopsies and/or hair follicles will be collected to establish cell lines. Investigators will ask all individuals providing samples to agree to potential future whole-genome sequencing in order to be able to potentially evaluate for genetic modifiers of these diseases.

These materials will be stored at a central repository (Greenwood Genetics Laboratory). The main purpose of these samples is to serve as durable materials for future analyses, however, a set of defined analyses will be performed on all samples. For the samples collected in the Rett syndrome cohort, investigators will perform X-chromosome inactivation studies and evaluate common polymorphisms in Brain derived neurotrophic factor (BDNF) and determine the contribution of these known factors to disease severity. For MECP2 Dup cohort investigators will characterize inflammatory markers in the plasma and correlate these with clinical features. Also for MECP2 Dup cohort investigators will perform detailed genomic breakpoint and gene content analysis and correlate this with disease severity. Similar analysis of genomic breakpoints and gene content will be performed on people with FOXG1 Duplications. Finally, in a pilot study, investigators will perform metabolic profiling on people from all disorders and evaluate for metabolic features correlated with disease severity, and metabolic features common or unique between these disorders. This work will provide a durable resource for future analysis, extend understanding of genotype/phenotype correlations, identify other biological factors contributing to disease severity, as well as provide the framework for the development of biomarkers of disease state and severity.

ELIGIBILITY:
Inclusion Criteria:

* Individuals of both genders and of all ages, with RTT, MECP2 Dup, and, RTT-related disorders including those with mutations or deletions in CDKL5 and FOXG1 genes, or those with RTT (atypical or typical) who are mutation negative. Additionally, unaffected family members of those people who meet the disease specific criteria stated will eligible.

Exclusion Criteria:

* Individuals who do not meet the above criteria will be excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Females and males of all ages must have complete testing for MECP2, FOXG1, and CDKL5 genes mutations AND must meet these requirements:
  Gene positive for a sequence mutation, duplication or deletion in one of these 3 genes.
  OR Meet consensus criteria for Rett syndrome (typical or atypical)
Sampling Method: Probability Sample
Enrollment: 752 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
X-chromosome inactivation in Rett syndrome (RTT) | 5 years
  Characterize X-chromosome inactivation in RTT and correlate with clinical severity.
Bdnf polymorphisms in RTT | 5 years
  Characterize Bdnf polymorphisms in RTT and correlate with clinical severity.
Inflammation markers in MECP2 duplication syndrome | 5 years
  Evaluate inflammation markers in MECP2 duplication syndrome and correlate with disease severity.
Biobanking of blood for Rett syndrome (RTT), MECP2 duplication syndrome, FOXG1, CDKL5, and MECP2 mutations not producing RTT | 5 years
  Blood will be collected and stored from participants with RTT, MECP2 duplication, FOXG1, CDKL5, and MECP2 mutations without RTT to analyze factors noted in Outcomes 1-3 and in secondary outcome 5 to correlate with disease severity.

SECONDARY OUTCOMES:
Breakpoints and gene content of MECP2 and FOXG1 duplications | 5 years
  Characterize breakpoints and gene content of MECP2 and FOXG1 duplications and correlate with disease severity

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey L Neul, MD, PhD, Study Chair — UCSD
Locations (12):
- United States (12):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - UCSF Benioff Children's Hospital Oakland, Oakland, California
  - University of California San Diego, San Diego, California
  - University of Colorado Denver, Denver, Colorado
  - Rush University Medical Center, Chicago, Illinois
  - Children's Hospital Boston, Boston, Massachusetts
  - Gillette Children's Specialty Healthcare, Minneapolis, Minnesota
  - Washington University School of Medicine and St. Louis Children's Hospital, St Louis, Missouri
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Greenwood Genetic Center, Greenwood, South Carolina
  - Vanderbilt University, Nashville, Tennessee
  - Baylor College of Medicine, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
The data sharing agreement approved by the Rare Disease Clinical Research Network will be employed.

REFERENCES:
- [Background] Hagberg B, Aicardi J, Dias K, Ramos O. A progressive syndrome of autism, dementia, ataxia, and loss of purposeful hand use in girls: Rett's syndrome: report of 35 cases. Ann Neurol. 1983 Oct;14(4):471-9. doi: 10.1002/ana.410140412. PMID 6638958
- [Background] Neul JL, Kaufmann WE, Glaze DG, Christodoulou J, Clarke AJ, Bahi-Buisson N, Leonard H, Bailey ME, Schanen NC, Zappella M, Renieri A, Huppke P, Percy AK; RettSearch Consortium. Rett syndrome: revised diagnostic criteria and nomenclature. Ann Neurol. 2010 Dec;68(6):944-50. doi: 10.1002/ana.22124. PMID 21154482
- [Background] Neul JL, Fang P, Barrish J, Lane J, Caeg EB, Smith EO, Zoghbi H, Percy A, Glaze DG. Specific mutations in methyl-CpG-binding protein 2 confer different severity in Rett syndrome. Neurology. 2008 Apr 15;70(16):1313-21. doi: 10.1212/01.wnl.0000291011.54508.aa. Epub 2008 Mar 12. PMID 18337588
- [Background] Nan X, Bird A. The biological functions of the methyl-CpG-binding protein MeCP2 and its implication in Rett syndrome. Brain Dev. 2001 Dec;23 Suppl 1:S32-7. doi: 10.1016/s0387-7604(01)00333-3. PMID 11738839
- [Background] Amir RE, Van den Veyver IB, Wan M, Tran CQ, Francke U, Zoghbi HY. Rett syndrome is caused by mutations in X-linked MECP2, encoding methyl-CpG-binding protein 2. Nat Genet. 1999 Oct;23(2):185-8. doi: 10.1038/13810. PMID 10508514
- [Background] Wan M, Lee SS, Zhang X, Houwink-Manville I, Song HR, Amir RE, Budden S, Naidu S, Pereira JL, Lo IF, Zoghbi HY, Schanen NC, Francke U. Rett syndrome and beyond: recurrent spontaneous and familial MECP2 mutations at CpG hotspots. Am J Hum Genet. 1999 Dec;65(6):1520-9. doi: 10.1086/302690. PMID 10577905
- [Background] Suter B, Treadwell-Deering D, Zoghbi HY, Glaze DG, Neul JL. Brief report: MECP2 mutations in people without Rett syndrome. J Autism Dev Disord. 2014 Mar;44(3):703-11. doi: 10.1007/s10803-013-1902-z. PMID 23921973
- [Background] Laurvick CL, de Klerk N, Bower C, Christodoulou J, Ravine D, Ellaway C, Williamson S, Leonard H. Rett syndrome in Australia: a review of the epidemiology. J Pediatr. 2006 Mar;148(3):347-52. doi: 10.1016/j.jpeds.2005.10.037. PMID 16615965
- [Background] Kerr AM, Armstrong DD, Prescott RJ, Doyle D, Kearney DL. Rett syndrome: analysis of deaths in the British survey. Eur Child Adolesc Psychiatry. 1997;6 Suppl 1:71-4. PMID 9452925
- [Background] Kirby RS, Lane JB, Childers J, Skinner SA, Annese F, Barrish JO, Glaze DG, Macleod P, Percy AK. Longevity in Rett syndrome: analysis of the North American Database. J Pediatr. 2010 Jan;156(1):135-138.e1. doi: 10.1016/j.jpeds.2009.07.015. PMID 19772971
- [Background] Guy J, Gan J, Selfridge J, Cobb S, Bird A. Reversal of neurological defects in a mouse model of Rett syndrome. Science. 2007 Feb 23;315(5815):1143-7. doi: 10.1126/science.1138389. Epub 2007 Feb 8. PMID 17289941
- [Background] Garg SK, Lioy DT, Cheval H, McGann JC, Bissonnette JM, Murtha MJ, Foust KD, Kaspar BK, Bird A, Mandel G. Systemic delivery of MeCP2 rescues behavioral and cellular deficits in female mouse models of Rett syndrome. J Neurosci. 2013 Aug 21;33(34):13612-20. doi: 10.1523/JNEUROSCI.1854-13.2013. PMID 23966684
- [Background] Chang Q, Khare G, Dani V, Nelson S, Jaenisch R. The disease progression of Mecp2 mutant mice is affected by the level of BDNF expression. Neuron. 2006 Feb 2;49(3):341-8. doi: 10.1016/j.neuron.2005.12.027. PMID 16446138
- [Background] Tropea D, Giacometti E, Wilson NR, Beard C, McCurry C, Fu DD, Flannery R, Jaenisch R, Sur M. Partial reversal of Rett Syndrome-like symptoms in MeCP2 mutant mice. Proc Natl Acad Sci U S A. 2009 Feb 10;106(6):2029-34. doi: 10.1073/pnas.0812394106. PMID 19208815
- [Background] Archer H, Evans J, Leonard H, Colvin L, Ravine D, Christodoulou J, Williamson S, Charman T, Bailey ME, Sampson J, de Klerk N, Clarke A. Correlation between clinical severity in patients with Rett syndrome with a p.R168X or p.T158M MECP2 mutation, and the direction and degree of skewing of X-chromosome inactivation. J Med Genet. 2007 Feb;44(2):148-52. doi: 10.1136/jmg.2006.045260. Epub 2006 Aug 11. PMID 16905679
- [Background] Leonard H, Bower C. Is the girl with Rett syndrome normal at birth? Dev Med Child Neurol. 1998 Feb;40(2):115-21. PMID 9489500
- [Background] Kerr AM. Early clinical signs in the Rett disorder. Neuropediatrics. 1995 Apr;26(2):67-71. doi: 10.1055/s-2007-979725. PMID 7566455
- [Background] Einspieler C, Kerr AM, Prechtl HF. Abnormal general movements in girls with Rett disorder: the first four months of life. Brain Dev. 2005 Nov;27 Suppl 1:S8-S13. doi: 10.1016/j.braindev.2005.03.014. Epub 2005 Sep 21. PMID 16182501
- [Background] Einspieler C, Kerr AM, Prechtl HF. Is the early development of girls with Rett disorder really normal? Pediatr Res. 2005 May;57(5 Pt 1):696-700. doi: 10.1203/01.PDR.0000155945.94249.0A. Epub 2005 Feb 17. PMID 15718369
- [Background] Downs J, Bebbington A, Kaufmann WE, Leonard H. Longitudinal hand function in Rett syndrome. J Child Neurol. 2011 Mar;26(3):334-40. doi: 10.1177/0883073810381920. Epub 2010 Oct 4. PMID 20921565
- [Background] Downs JA, Bebbington A, Jacoby P, Msall ME, McIlroy O, Fyfe S, Bahi-Buisson N, Kaufmann WE, Leonard H. Gross motor profile in rett syndrome as determined by video analysis. Neuropediatrics. 2008 Aug;39(4):205-10. doi: 10.1055/s-0028-1104575. Epub 2009 Jan 22. PMID 19165708
- [Background] Neul, J.L. Rett Syndrome and MECP2-Related Disorders. in Autism Spectrum Disorders (eds. Amaral, D., Geschwind, D. & Dawson, G.) 776-800 (Oxford University Press, New York, 2011).
- [Background] Nectoux J, Bahi-Buisson N, Guellec I, Coste J, De Roux N, Rosas H, Tardieu M, Chelly J, Bienvenu T. The p.Val66Met polymorphism in the BDNF gene protects against early seizures in Rett syndrome. Neurology. 2008 May 27;70(22 Pt 2):2145-51. doi: 10.1212/01.wnl.0000304086.75913.b2. Epub 2008 Apr 23. PMID 18434641
- [Background] Zeev BB, Bebbington A, Ho G, Leonard H, de Klerk N, Gak E, Vecsler M, Christodoulou J. The common BDNF polymorphism may be a modifier of disease severity in Rett syndrome. Neurology. 2009 Apr 7;72(14):1242-7. doi: 10.1212/01.wnl.0000345664.72220.6a. PMID 19349604
- [Background] Egan MF, Kojima M, Callicott JH, Goldberg TE, Kolachana BS, Bertolino A, Zaitsev E, Gold B, Goldman D, Dean M, Lu B, Weinberger DR. The BDNF val66met polymorphism affects activity-dependent secretion of BDNF and human memory and hippocampal function. Cell. 2003 Jan 24;112(2):257-69. doi: 10.1016/s0092-8674(03)00035-7. PMID 12553913
- [Background] Buchovecky CM, Turley SD, Brown HM, Kyle SM, McDonald JG, Liu B, Pieper AA, Huang W, Katz DM, Russell DW, Shendure J, Justice MJ. A suppressor screen in Mecp2 mutant mice implicates cholesterol metabolism in Rett syndrome. Nat Genet. 2013 Sep;45(9):1013-20. doi: 10.1038/ng.2714. Epub 2013 Jul 28. PMID 23892605
- [Background] Bebbington A, Anderson A, Ravine D, Fyfe S, Pineda M, de Klerk N, Ben-Zeev B, Yatawara N, Percy A, Kaufmann WE, Leonard H. Investigating genotype-phenotype relationships in Rett syndrome using an international data set. Neurology. 2008 Mar 11;70(11):868-75. doi: 10.1212/01.wnl.0000304752.50773.ec. PMID 18332345
- [Background] Ramocki MB, Peters SU, Tavyev YJ, Zhang F, Carvalho CM, Schaaf CP, Richman R, Fang P, Glaze DG, Lupski JR, Zoghbi HY. Autism and other neuropsychiatric symptoms are prevalent in individuals with MeCP2 duplication syndrome. Ann Neurol. 2009 Dec;66(6):771-82. doi: 10.1002/ana.21715. PMID 20035514
- [Background] Peters SU, Hundley RJ, Wilson AK, Carvalho CM, Lupski JR, Ramocki MB. Brief report: regression timing and associated features in MECP2 duplication syndrome. J Autism Dev Disord. 2013 Oct;43(10):2484-90. doi: 10.1007/s10803-013-1796-9. PMID 23456562
- [Background] Friez MJ, Jones JR, Clarkson K, Lubs H, Abuelo D, Bier JA, Pai S, Simensen R, Williams C, Giampietro PF, Schwartz CE, Stevenson RE. Recurrent infections, hypotonia, and mental retardation caused by duplication of MECP2 and adjacent region in Xq28. Pediatrics. 2006 Dec;118(6):e1687-95. doi: 10.1542/peds.2006-0395. Epub 2006 Nov 6. PMID 17088400
- [Background] Van Esch H, Bauters M, Ignatius J, Jansen M, Raynaud M, Hollanders K, Lugtenberg D, Bienvenu T, Jensen LR, Gecz J, Moraine C, Marynen P, Fryns JP, Froyen G. Duplication of the MECP2 region is a frequent cause of severe mental retardation and progressive neurological symptoms in males. Am J Hum Genet. 2005 Sep;77(3):442-53. doi: 10.1086/444549. Epub 2005 Jul 29. PMID 16080119
- [Background] Ramocki MB, Tavyev YJ, Peters SU. The MECP2 duplication syndrome. Am J Med Genet A. 2010 May;152A(5):1079-88. doi: 10.1002/ajmg.a.33184. PMID 20425814
- [Background] Van Esch H. MECP2 Duplication Syndrome. Mol Syndromol. 2012 Apr;2(3-5):128-136. doi: 10.1159/000329580. Epub 2011 Jul 5. PMID 22679399
- [Background] Carvalho CM, Ramocki MB, Pehlivan D, Franco LM, Gonzaga-Jauregui C, Fang P, McCall A, Pivnick EK, Hines-Dowell S, Seaver LH, Friehling L, Lee S, Smith R, Del Gaudio D, Withers M, Liu P, Cheung SW, Belmont JW, Zoghbi HY, Hastings PJ, Lupski JR. Inverted genomic segments and complex triplication rearrangements are mediated by inverted repeats in the human genome. Nat Genet. 2011 Oct 2;43(11):1074-81. doi: 10.1038/ng.944. PMID 21964572
- [Background] Yang T, Ramocki MB, Neul JL, Lu W, Roberts L, Knight J, Ward CS, Zoghbi HY, Kheradmand F, Corry DB. Overexpression of methyl-CpG binding protein 2 impairs T(H)1 responses. Sci Transl Med. 2012 Dec 5;4(163):163ra158. doi: 10.1126/scitranslmed.3004430. PMID 23220634
- [Background] Na ES, Nelson ED, Adachi M, Autry AE, Mahgoub MA, Kavalali ET, Monteggia LM. A mouse model for MeCP2 duplication syndrome: MeCP2 overexpression impairs learning and memory and synaptic transmission. J Neurosci. 2012 Feb 29;32(9):3109-17. doi: 10.1523/JNEUROSCI.6000-11.2012. PMID 22378884
- [Background] Na ES, Nelson ED, Kavalali ET, Monteggia LM. The impact of MeCP2 loss- or gain-of-function on synaptic plasticity. Neuropsychopharmacology. 2013 Jan;38(1):212-9. doi: 10.1038/npp.2012.116. Epub 2012 Jul 11. PMID 22781840
- [Background] Ariani F, Mari F, Pescucci C, Longo I, Bruttini M, Meloni I, Hayek G, Rocchi R, Zappella M, Renieri A. Real-time quantitative PCR as a routine method for screening large rearrangements in Rett syndrome: Report of one case of MECP2 deletion and one case of MECP2 duplication. Hum Mutat. 2004 Aug;24(2):172-7. doi: 10.1002/humu.20065. PMID 15241799
- [Background] Meins M, Lehmann J, Gerresheim F, Herchenbach J, Hagedorn M, Hameister K, Epplen JT. Submicroscopic duplication in Xq28 causes increased expression of the MECP2 gene in a boy with severe mental retardation and features of Rett syndrome. J Med Genet. 2005 Feb;42(2):e12. doi: 10.1136/jmg.2004.023804. No abstract available. PMID 15689435
- [Background] Grasshoff U, Bonin M, Goehring I, Ekici A, Dufke A, Cremer K, Wagner N, Rossier E, Jauch A, Walter M, Bauer C, Bauer P, Horber K, Beck-Woedl S, Wieczorek D. De novo MECP2 duplication in two females with random X-inactivation and moderate mental retardation. Eur J Hum Genet. 2011 May;19(5):507-12. doi: 10.1038/ejhg.2010.226. Epub 2011 Feb 16. PMID 21326285
- [Background] del Gaudio D, Fang P, Scaglia F, Ward PA, Craigen WJ, Glaze DG, Neul JL, Patel A, Lee JA, Irons M, Berry SA, Pursley AA, Grebe TA, Freedenberg D, Martin RA, Hsich GE, Khera JR, Friedman NR, Zoghbi HY, Eng CM, Lupski JR, Beaudet AL, Cheung SW, Roa BB. Increased MECP2 gene copy number as the result of genomic duplication in neurodevelopmentally delayed males. Genet Med. 2006 Dec;8(12):784-92. doi: 10.1097/01.gim.0000250502.28516.3c. PMID 17172942
- [Background] Carvalho CM, Zhang F, Liu P, Patel A, Sahoo T, Bacino CA, Shaw C, Peacock S, Pursley A, Tavyev YJ, Ramocki MB, Nawara M, Obersztyn E, Vianna-Morgante AM, Stankiewicz P, Zoghbi HY, Cheung SW, Lupski JR. Complex rearrangements in patients with duplications of MECP2 can occur by fork stalling and template switching. Hum Mol Genet. 2009 Jun 15;18(12):2188-203. doi: 10.1093/hmg/ddp151. Epub 2009 Mar 26. PMID 19324899
- [Background] Reardon W, Donoghue V, Murphy AM, King MD, Mayne PD, Horn N, Birk Moller L. Progressive cerebellar degenerative changes in the severe mental retardation syndrome caused by duplication of MECP2 and adjacent loci on Xq28. Eur J Pediatr. 2010 Aug;169(8):941-9. doi: 10.1007/s00431-010-1144-4. Epub 2010 Feb 23. PMID 20177701
- [Background] Honda S, Hayashi S, Nakane T, Imoto I, Kurosawa K, Mizuno S, Okamoto N, Kato M, Yoshihashi H, Kubota T, Nakagawa E, Goto Y, Inazawa J. The incidence of hypoplasia of the corpus callosum in patients with dup (X)(q28) involving MECP2 is associated with the location of distal breakpoints. Am J Med Genet A. 2012 Jun;158A(6):1292-303. doi: 10.1002/ajmg.a.35321. Epub 2012 Apr 23. PMID 22528406
- [Background] Vignoli A, Borgatti R, Peron A, Zucca C, Ballarati L, Bonaglia C, Bellini M, Giordano L, Romaniello R, Bedeschi MF, Epifanio R, Russo S, Caselli R, Giardino D, Darra F, La Briola F, Banderali G, Canevini MP. Electroclinical pattern in MECP2 duplication syndrome: eight new reported cases and review of literature. Epilepsia. 2012 Jul;53(7):1146-55. doi: 10.1111/j.1528-1167.2012.03501.x. Epub 2012 May 11. PMID 22578097
- [Background] Lupski JR. Genomic disorders ten years on. Genome Med. 2009 Apr 24;1(4):42. doi: 10.1186/gm42. PMID 19439022
- [Background] Hanashima C, Fernandes M, Hebert JM, Fishell G. The role of Foxg1 and dorsal midline signaling in the generation of Cajal-Retzius subtypes. J Neurosci. 2007 Oct 10;27(41):11103-11. doi: 10.1523/JNEUROSCI.1066-07.2007. PMID 17928452
- [Background] Brancaccio M, Pivetta C, Granzotto M, Filippis C, Mallamaci A. Emx2 and Foxg1 inhibit gliogenesis and promote neuronogenesis. Stem Cells. 2010 Jul;28(7):1206-18. doi: 10.1002/stem.443. PMID 20506244
- [Background] Bahi-Buisson N, Villeneuve N, Caietta E, Jacquette A, Maurey H, Matthijs G, Van Esch H, Delahaye A, Moncla A, Milh M, Zufferey F, Diebold B, Bienvenu T. Recurrent mutations in the CDKL5 gene: genotype-phenotype relationships. Am J Med Genet A. 2012 Jul;158A(7):1612-9. doi: 10.1002/ajmg.a.35401. Epub 2012 Jun 7. PMID 22678952
- [Background] Nemos C, Lambert L, Giuliano F, Doray B, Roubertie A, Goldenberg A, Delobel B, Layet V, N'guyen MA, Saunier A, Verneau F, Jonveaux P, Philippe C. Mutational spectrum of CDKL5 in early-onset encephalopathies: a study of a large collection of French patients and review of the literature. Clin Genet. 2009 Oct;76(4):357-71. doi: 10.1111/j.1399-0004.2009.01194.x. PMID 19793311
- [Background] Brunetti-Pierri N, Paciorkowski AR, Ciccone R, Della Mina E, Bonaglia MC, Borgatti R, Schaaf CP, Sutton VR, Xia Z, Jelluma N, Ruivenkamp C, Bertrand M, de Ravel TJ, Jayakar P, Belli S, Rocchetti K, Pantaleoni C, D'Arrigo S, Hughes J, Cheung SW, Zuffardi O, Stankiewicz P. Duplications of FOXG1 in 14q12 are associated with developmental epilepsy, mental retardation, and severe speech impairment. Eur J Hum Genet. 2011 Jan;19(1):102-7. doi: 10.1038/ejhg.2010.142. Epub 2010 Aug 25. PMID 20736978
- [Background] Wang IT, Allen M, Goffin D, Zhu X, Fairless AH, Brodkin ES, Siegel SJ, Marsh ED, Blendy JA, Zhou Z. Loss of CDKL5 disrupts kinome profile and event-related potentials leading to autistic-like phenotypes in mice. Proc Natl Acad Sci U S A. 2012 Dec 26;109(52):21516-21. doi: 10.1073/pnas.1216988110. Epub 2012 Dec 10. PMID 23236174
- [Background] Huppke P, Held M, Laccone F, Hanefeld F. The spectrum of phenotypes in females with Rett Syndrome. Brain Dev. 2003 Aug;25(5):346-51. doi: 10.1016/s0387-7604(03)00018-4. PMID 12850514
- [Background] Rajaei S, Erlandson A, Kyllerman M, Albage M, Lundstrom I, Karrstedt EL, Hagberg B. Early infantile onset ''congenital'' Rett syndrome variants: Swedish experience through four decades and mutation analysis. J Child Neurol. 2011 Jan;26(1):65-71. doi: 10.1177/0883073810374125. PMID 21212452
- [Background] Nectoux J, Fichou Y, Cagnard N, Bahi-Buisson N, Nusbaum P, Letourneur F, Chelly J, Bienvenu T. Cell cloning-based transcriptome analysis in cyclin-dependent kinase-like 5 mutation patients with severe epileptic encephalopathy. J Mol Med (Berl). 2011 Feb;89(2):193-202. doi: 10.1007/s00109-010-0699-x. Epub 2010 Nov 24. PMID 21107515
- [Background] Ricciardi S, Kilstrup-Nielsen C, Bienvenu T, Jacquette A, Landsberger N, Broccoli V. CDKL5 influences RNA splicing activity by its association to the nuclear speckle molecular machinery. Hum Mol Genet. 2009 Dec 1;18(23):4590-602. doi: 10.1093/hmg/ddp426. Epub 2009 Sep 9. PMID 19740913
- [Background] Weaving LS, Christodoulou J, Williamson SL, Friend KL, McKenzie OL, Archer H, Evans J, Clarke A, Pelka GJ, Tam PP, Watson C, Lahooti H, Ellaway CJ, Bennetts B, Leonard H, Gecz J. Mutations of CDKL5 cause a severe neurodevelopmental disorder with infantile spasms and mental retardation. Am J Hum Genet. 2004 Dec;75(6):1079-93. doi: 10.1086/426462. Epub 2004 Oct 18. PMID 15492925
- [Background] Bahi-Buisson N, Kaminska A, Boddaert N, Rio M, Afenjar A, Gerard M, Giuliano F, Motte J, Heron D, Morel MA, Plouin P, Richelme C, des Portes V, Dulac O, Philippe C, Chiron C, Nabbout R, Bienvenu T. The three stages of epilepsy in patients with CDKL5 mutations. Epilepsia. 2008 Jun;49(6):1027-37. doi: 10.1111/j.1528-1167.2007.01520.x. Epub 2008 Feb 7. PMID 18266744
- [Background] Bahi-Buisson N, Nectoux J, Rosas-Vargas H, Milh M, Boddaert N, Girard B, Cances C, Ville D, Afenjar A, Rio M, Heron D, N'guyen Morel MA, Arzimanoglou A, Philippe C, Jonveaux P, Chelly J, Bienvenu T. Key clinical features to identify girls with CDKL5 mutations. Brain. 2008 Oct;131(Pt 10):2647-61. doi: 10.1093/brain/awn197. Epub 2008 Sep 12. PMID 18790821
- [Background] Fehr S, Wilson M, Downs J, Williams S, Murgia A, Sartori S, Vecchi M, Ho G, Polli R, Psoni S, Bao X, de Klerk N, Leonard H, Christodoulou J. The CDKL5 disorder is an independent clinical entity associated with early-onset encephalopathy. Eur J Hum Genet. 2013 Mar;21(3):266-73. doi: 10.1038/ejhg.2012.156. Epub 2012 Aug 8. PMID 22872100
- [Background] Melani F, Mei D, Pisano T, Savasta S, Franzoni E, Ferrari AR, Marini C, Guerrini R. CDKL5 gene-related epileptic encephalopathy: electroclinical findings in the first year of life. Dev Med Child Neurol. 2011 Apr;53(4):354-60. doi: 10.1111/j.1469-8749.2010.03889.x. Epub 2011 Feb 11. PMID 21309761
- [Background] Elia M, Falco M, Ferri R, Spalletta A, Bottitta M, Calabrese G, Carotenuto M, Musumeci SA, Lo Giudice M, Fichera M. CDKL5 mutations in boys with severe encephalopathy and early-onset intractable epilepsy. Neurology. 2008 Sep 23;71(13):997-9. doi: 10.1212/01.wnl.0000326592.37105.88. PMID 18809835
- See also: International Rett Syndrome Foundation website — http://www.rettsyndrome.org/